CLINICAL TRIAL: NCT07384975
Title: A Phase 2a, Multicenter, Randomized, Double-blind, Placebo-controlled Study of NAV-240 in Adult Participants With Moderate-to-Severe Hidradenitis Suppurativa
Brief Title: A Study to Assess NAV-240 in Adult Participants With Hidradenitis Suppurativa
Acronym: Mainsail
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navigator Medicines, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAV-240-201; 2025-523557-33-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa (HS)
Keywords: NAV-240; HS; Hidradenitis Suppurativa; Phase 2; Moderate-to-Severe HS
MeSH Terms: conditions — Hidradenitis Suppurativa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NAV-240 Dose 1 (Experimental): NAV-240 Dose 1
  Interventions: Drug: NAV-240
- NAV-240 Dose 2 (Experimental): NAV-240 Dose 2
  Interventions: Drug: NAV-240
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo to match NAV-240

INTERVENTIONS:
Drug: NAV-240 — NAV-240 for Intravenous Infusion
  Arms: NAV-240 Dose 1; NAV-240 Dose 2
Drug: Placebo to match NAV-240 — Placebo to match NAV-240 for Intravenous Infusion
  Arms: Placebo

SUMMARY:
The main objective of this study is to determine if NAV-240 works more effectively than a dummy treatment (placebo) for participants with moderate-to-severe HS. The main endpoint of this study is the percentage of participants achieving Hidradenitis Suppurativa Clinical Response (HiSCR) 75 at Week 16, meaning at least a 75% reduction in inflamed skin bumps (abscess and inflammatory nodule (AN) count) with no increase in number of abscesses or draining tunnels (channels under the skin that leak fluid or pus) compared to the baseline (start of the study).

Participants will:

* Receive NAV-240 dose 1, NAV-240 dose 2 or placebo as a drip into the veins (intravenous infusion).
* Visit the clinic up to 9 times for checkups and tests over 22 weeks.
* Complete a daily diary about their skin pain.

ELIGIBILITY:
Inclusion Criteria:

* History of HS for ≥ 6 months
* Abscesses and Inflammatory Nodules (lesion) count ≥ 5
* Inflammatory HS lesions in at least 2 different body regions, one of which must be Hurley Stage II or III
* Inadequate response to at least one course of antibiotics
* Topical antiseptics are not required but allowed. If in use, the participant must agree to use one single product consistently through Week 16.
* Use of oral antibiotics is allowed during the study under the following conditions: the dose and regimen must remain stable until Week 16. Allowed oral antibiotics include doxycycline, minocycline, or tetracycline.
* Female participants of childbearing potential must have a negative pregnancy test
* Participants of reproductive potential must use a highly effective method of contraception

Exclusion Criteria:

* > 20 draining tunnel count
* Active skin disease (bacterial, fungal, viral infection) that, in the opinion of the Investigator, could interfere with assessment of HS or requires treatment with antibiotic(s) also used to treat HS.
* Has had major surgery, including HS surgery, within 12 weeks prior to Day 1
* History of alcohol or drug abuse within the past 2 years.
* A positive urine drug screen at Screening
* History or evidence of human immunodeficiency virus (HIV), hepatitis B or hepatitis C virus (HCV), or a positive test at Screening
* History or current diagnosis of active tuberculosis (TB), untreated latent TB infection (LTBI), or undergoing current treatment for LTBI, determined by positive TB test
* History of moderate to severe heart failure or recent (within past 6 months) cerebrovascular accident, myocardial infarction, or coronary stenting.
* History of immune deficiency

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving Hidradenitis Suppurativa Clinical Response (HiSCR) 75 | Baseline to Week 16
  HiSCR75 is defined as at least a 75% reduction in total abscess and inflammatory nodule count (AN count) with no increase in abscess count and no increase in draining tunnel count relative to baseline.

SECONDARY OUTCOMES:
Proportion of participants achieving skin pain numeric rating scale (NRS) 30 response | Baseline to Week 16
  NRS30 is defined as a ≥ 30% reduction and at least a 2-unit reduction from baseline in skin pain on the NRS, for participants with a baseline skin pain NRS ≥ 3, based on the weekly average of the worst skin pain in a 24-hour recall period (maximal daily pain).
Proportion of participants achieving HiSCR50 | Baseline to Week 16
  HiSCR50 is defined as at least a 50% reduction in total AN count with no increase in abscess count and no increase in draining tunnel count relative to baseline.
Proportion of participants achieving a Dermatology Life Quality Index (DLQI) improvement (reduction) of ≥ 4 points among participants with DLQI ≥ 4 at baseline | Baseline to Week 16
Proportion of participants with HS flare | Baseline to Week 16
Change in the International Hidradenitis Suppurativa Severity Score System (IHS4) scores | Baseline to Week 16
Change from baseline in AN count | Baseline to Week 16
Change from baseline in the number of draining tunnels | Baseline to Week 16

OTHER OUTCOMES:
Incidence of TEAEs, SAEs and adverse events of special interest (AESIs) | Baseline to Week 16

CONTACTS AND LOCATIONS:
Overall Officials: Lara Pupim, MD, MSCI, Study Director — Navigator Medicines, Inc.
Locations (10):
- United States (10):
  - Medical Dermatology Specialist, Phoenix, Arizona
  - Accel Research Sites Network, Maitland, Florida
  - Floridian Research Institute, Miami, Florida
  - Cordova Research Institute, Miami, Florida
  - Tory Sullivan MD PA - Dermatology, North Miami Beach, Florida
  - MplusM - D&H Tamarac Research Center, Tamarac, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Kentucky Advanced Medical Research LLC, Murray, Kentucky
  - ActivMed Practices & Research, LLC, Portsmouth, New Hampshire
  - Equity Medical, LLC, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No